CLINICAL TRIAL: NCT03350438
Title: Participation in Everyday Occupations and Perception of Quality of Life-comparing Adults Eith PTSD With Typical Adults and Assessing the Relationship Between the Two Measures
Brief Title: Participation in Occupations and Perception of Quality of Life, Comparing Adults With and Without PTSD
Acronym: PTSD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0023-17-ziv
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: participation; quality of life; occupational therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTSD Patients: patients ranging 18-60, diagnosed with PTSD following a trauma that occured over one year before the current study and do not have other health problems that may affect their everyday participation.
- healthy adults: healthy adults, ranging 18-60, without any health problems that may affect their everyday participation.

SUMMARY:
This study assesses the relationship between participation and quality of life the way adults with and without Post Traumatic Stress Disorder (PTSD) experience it in everyday life. Both groups will fill out Questionnaires and the answers will be compared. In addition different aspects of dissociation will be taken in to consideration.

DETAILED DESCRIPTION:
Post Traumatic Stress Disorder has been known to severely impair participation in everyday activities such as work, recreation and social participation. In turn, these impairments can diminish quality of life. However, the relationship between PTSD, functioning and quality of life remains incompletely understood.

Since achieving full participation in daily activities is the main goal of occupational therapy, and since quality of life is a primary treatment success measure, it is important to fully understand the relationship between PTSD, participation and quality of life.

Various studies show that dissociation affects different body functions that manage and monitor mental functioning. Since quality of life is a subjective measure that relies on one's ability to mentally represent himself and others it is important to tack into consideration the way that dissociation affects the relationships described above.

The research contains 4 Questionnaires that will be filed out by the participants and the data from the Questionnaires will be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking, read and write in Hebrew, have been diagnosed with PTSD following a trauma that occurred over one year before the current study.

Exclusion Criteria:

* Other psychiatric disorders, cognitive or physical impairments.

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: men, age 18-60, Hebrew speaking, read and write in Hebrew, have been diagnosed with PTSD following a trauma that occurred over one year before the current study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
self reported quality of life | two weeks
  self reported quality of life, 26 items scored 1-5 (1=not at all/very bad 5=very much/very good) regarding how a person feels about his quality of life, health and other aspects of life in the past two weeks.

SECONDARY OUTCOMES:
Self Reported Dissociation | 24-48 hours
  Self Reported Dissociative Experiences, 10 items scored 1-5 (1=not at all true 5=always true) regarding different experiences and reactions during the traumatic event and after.
self reported participation | 1 month
  88 different activities that are rated 0-1 in comparison to before the trauma. 0= if the person is not currently participating 0.5= if the person is participating less then before the trauma 1= if the person is participating the same as before the trauma
self reported ptsd symptoms | 1 month
  self reported ptsd symptoms, 17 items scored 0-3, regarding different reactions, feelings and experiences according to what the patient has experienced in the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Isakson, PHD, Principal Investigator — Ziv Hospital
Locations (1):
- Ziv Hospital, Safed, Galilee, Israel